CLINICAL TRIAL: NCT03394846
Title: Testing Products to Increase Children's Physical Activity in the Classroom: Identifying What Works and What Doesn't
Brief Title: Classroom Activities
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, R. Glenn Weaver, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00069012
Record Dates: First submitted 2017-11-10; First posted 2018-01-09 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of Existing MI Products (Experimental): We will test the impact of three widely available MI products (GoNoodle, Take10, ABC for Fitness) on students' physical activity with 60 elementary classroom teachers.
  Interventions: Behavioral: Test of Existing MI Products

INTERVENTIONS:
Behavioral: Test of Existing MI Products — Three widely available MI products (GoNoodle, Take10, ABC for Fitness) will be tested by teachers in their classrooms. Teachers will participate in the study for four weeks (one baseline week, one week for each product).

SUMMARY:
Movement integration programs that incorporate physical activity into academics are widely available for teachers to use, and have been shown to provide meaningful amounts of physical activity, improve on-task behavior, enhance cognitive function, and increase standardized test scores of children. However, teachers rarely use these programs. This project aims to use product testing and development methodologies to test current movement integration programs, identify critical attributes of those programs that hinder or enhance uptake by teachers, and develop a novel movement integration program based on those attributes.

DETAILED DESCRIPTION:
Movement integration (MI) is a strategy for integrating physical activity into general education classroom time. National organizations have identified MI as a key strategy for helping children accumulate the recommended 60 minutes of moderate-to-vigorous physical activity per day. Research has consistently demonstrated that MI can provide meaningful amounts of physical activity, improve on-task behavior, enhance cognitive function, and increase standardized test scores.This strategy is also increasingly important because children spend less and less time in active school settings, such as recess and physical education. However, teachers rarely incorporate MI into their classrooms.

In order to encourage teachers to use MI more regularly, it is essential to understand which MI product attributes lead to greater use. While some work has been done to identify which attributes of MI products enhance teacher use, this work has either examined the use of MI as a general concept (i.e., what would make teachers more likely to infuse physical activity [PA] into their classroom routines); or was conducted within the context of a single MI product (i.e., what makes teachers more likely to implement a specific MI product, such as Take 10).These approaches have two major limitations. First, studies that examined MI as a general concept (i.e., what would make teachers more likely to infuse physical activity into their classroom routines) are limited because teachers were not able to test MI products. Second, because previous studies solicited feedback on a single MI product, even though several MI products with varying attributes are available, teachers' ability to identify desirable MI product attributes across MI products was limited.

Currently, six MI products are widely available to teachers. These products differ significantly in their degree of (a) academic focus, (b) level of teacher involvement, and (c) time commitment for planning and implementation. For example, Go Noodle is a website that contains short (3-5 minute) videos of mostly non-academic MI activities. Teachers can simply select a video to play. Conversely, the Take 10 product consists of activity cards that present physical activities infused with academic content, plus instructions for how teachers can organize and implement the activities. These two products represent opposite ends of the MI product spectrum, but no one MI product includes all of the key attributes that may encourage use. Understanding the attributes that teachers want in MI products would allow researchers and educators to design products that have greater appeal and are more likely to be used (i.e., increased implementation).

Product testing is one way to identify attributes that enhance or hinder uptake by teachers. Product testing is the process of measuring the properties or performance of products. Two of the most common product testing techniques are in-home use tests, and discrete choice experiments (DCE). In-home use tests allow potential consumers (in this case teachers) to use a product as they normally would in their natural setting. DCEs involve asking individuals to identify their preferences when given a hypothetical set of attributes products could contain.Product testing is essential when developing new products, because it can help to produce superior products, by identifying critical attributes that consumers desire. Research has categorically shown that including consumers in the development of new products is critical to the success of the products. However, the process of developing previous MI products has not included this step.

This study will expand the evidence related to implementation of MI by classroom teachers by identifying product attributes that will lead to increased use of MI products by teachers. To do this we will draw upon product testing research techniques to test widely-available MI products and to identify attributes of MI products that make them more or less usable. We will accomplish the following specific aims:

Aim 1: Identify the key attributes of Movement Integration products that teachers prefer and do not prefer, using a DCE and in-class product testing.

Aim 2: Develop a prototype Movement Integration product that incorporates the critical attributes identified by teachers in Aim 1.

Aim 3: Conduct a pilot test of the prototype Movement Integration product developed in Aim 2 to evaluate teacher implementation, the product's effect on children's activity levels during classroom time, and cost.

This project is significant because MI can reach virtually all children each day at school. The project is innovative because it will produce a MI product prototype using product testing techniques with classroom teachers. The expected project outcome is a MI product prototype with the potential to be more widely implemented throughout the country.

Updates Due to Covid-19: Because of the closure of schools due to the novel SARS-CoV-2 (COVID-19) pandemic and due to the pilot data collected in Aim 1 the design of this study has undergone changes. Upon the completion of Aim 1 it became clear that existing MI products contained all of the key attributes that teachers desired. Thus, the decision was made not to create a novel MI product but rather to test the impact of the three products that teachers ranked the highest in Aim 1 on students' physical activity. Teachers began testing products in January of 2020 and all of the participating schools closed their doors in March of 2020 due to COVID-19. Prior to the closure teachers were able to complete a baseline week and test one product. These schools reopened in the fall of 2021 but have not allowed external visitors to the school, including study research teams. Thus it has been and remains impossible to complete the study as intended. Given that the grant funding for this project has come to a close it is the investigators' intention to publish the findings as is, while recognizing and transparently reporting their limitations.

ELIGIBILITY:
* Participants must be an elementary classroom teacher.
* Must be employed full time by their school district
* Must be the primary classroom teacher with a class of 15 or more students of elementary age

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We will not share IPD data.

REFERENCES:
- [Derived] Weaver RG, Dugger R, Burkart S, von Klinggraeff L, Hunt ET, Beets MW, Webster CA, Chen B, Armstrong B, Adams EL, Rehling J. Classroom teachers' "off-the-shelf" use of movement integration products and its impact on children's sedentary behavior and physical activity. Transl Behav Med. 2022 Dec 30;12(12):1116-1123. doi: 10.1093/tbm/ibac055. PMID 35998100

RESULTS

PARTICIPANT FLOW:
Groups:
- ABC for Fitness: ABC for Fitness is a free guidebook designed to provide teachers with ideas to intersperse physical activity bursts throughout the school day. Each activity burst has three components: A. Warm-up, B. Core Activity (e.g., exercise, stretching), and C. Cool Down lasting a maximum of five minutes. This resource contains academic content which teachers are encouraged to integrate into their lesson plans.
- Take 10: Take 10 is a classroom-based guidebook that provides teachers with grade-specific academic lessons that are integrated with PA. Each lesson offers an opportunity for the students to be physically active while learning academic content in one of five subject areas: language arts, math, science, social studies, or general health. Each activity is designed to last for a maximum of ten minutes. Take 10 employs a tiered pricing scheme based on grade level and ranges in cost from $85-$112.
- GoNoodle: GoNoodle is a free, online resource that contains a series of videos integrating grade-specific academic content with a variety of physical activities (e.g., dance, exercise, yoga) set to music and activity breaks. These activities are non-teacher led and incorporate elements of social and emotional wellness to support child development. Video length tends to run between 5-10 minutes. For a cost (i.e., $99 per year), GoNoodle Plus offers extended curricula videos, more learning games, and includes printable activities. Teachers were provided with the GoNoodle Plus version during product testing.
Period: Overall Study
Arm/Group | ABC for Fitness | Take 10 | GoNoodle
Started | 19 | 34 | 4
Completed | 19 | 34 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ABC for Fitness: One baseline week was followed by a week where teachers used ABC for Fitness. ABC for Fitness is a free guidebook designed to provide teachers with ideas to intersperse physical activity bursts throughout the school day. Each activity burst has three components: A. Warm-up, B. Core Activity (e.g., exercise, stretching), and C. Cool Down lasting a maximum of five minutes. This resource contains academic content which teachers are encouraged to integrate into their lesson plans. During the baseline week teachers were asked to go about their regularly scheduled classroom activities like any other typical week. During the intervention week teachers were allowed to determine the times and duration of product use and there were no restrictions or guidance from the research team. Teachers were informed that they were free to use any feature of the product to implement in their classroom as often or infrequently as they preferred. All teachers were informed of the study's purpose and that the study staff were not affiliated with the MI products.
- Take 10: One baseline week was followed by a week where teachers used Take 10. Take 10 is a classroom-based guidebook that provides teachers with grade-specific academic lessons that are integrated with PA. Each lesson offers an opportunity for the students to be physically active while learning academic content in one of five subject areas: language arts, math, science, social studies, or general health. Each activity is designed to last for a maximum of ten minutes. Take 10 employs a tiered pricing scheme based on grade level and ranges in cost from $85-$112.During the baseline week teachers were asked to go about their regularly scheduled classroom activities like any other typical week. During the intervention week teachers were allowed to determine the times and duration of product use and there were no restrictions or guidance from the research team. Teachers were informed that they were free to use any feature of the product to implement in their classroom as often or infrequently as they preferred. All teachers were informed of the study's purpose and that the study staff were not affiliated with the MI products.
- GoNoodle: One baseline week was followed by a week where teachers used GoNoodle. GoNoodle is a free, online resource that contains a series of videos integrating grade-specific academic content with a variety of physical activities (e.g., dance, exercise, yoga) set to music and activity breaks. These activities are non-teacher led and incorporate elements of social and emotional wellness to support child development. Video length tends to run between 5-10 minutes. For a cost (i.e., $99 per year), GoNoodle Plus offers extended curricula videos, more learning games, and includes printable activities. Teachers were provided with the GoNoodle Plus version during product testing. During the baseline week teachers were asked to go about their regularly scheduled classroom activities like any other typical week. During the intervention week teachers were allowed to determine the times and duration of product use and there were no restrictions or guidance from the research team. Teachers were informed that they were free to use any feature of the product to implement in their classroom as often or infrequently as they preferred. All teachers were informed of the study's purpose and that the study staff were not affiliated with the MI products.
- Total: Total of all reporting groups
Arm/Group | ABC for Fitness | Take 10 | GoNoodle | Total
Number analyzed (Participants) | 19 | 34 | 4 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (10.6) | 48.6 (5.9) | 39.8 (10.2) | 46.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 34 | 4 | 57
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 32 | 0 | 44
  White | 7 | 0 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 34 | 4 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in Use of Movement Integration Strategies (Mean Per Day)
Description: Change in self-reported use of movement integration strategies per day. Teachers will complete a weekly log of movement integration product implementation. To complete the log, each teacher will log onto a password-protected website. Teachers will indicate the number of MI product uses per day. If teachers fail to complete the log they will receive an email reminder.
Time Frame: 5 school days (Data was averaged across the 5 days) at baseline (teachers did not have the movement integration product) and outcome (one week following baseline when teachers were provided the movement integration product)
Measure: Mean (95% Confidence Interval); unit: Change in movement strategy use per day
Arm/Group | ABC for Fitness | Take 10 | GoNoodle
Number analyzed (Participants) | 19 | 34 | 4
Change in movement strategy use per day | 0.4 [-0.1 to 0.7] | 0.1 [-0.1 to 0.2] | 0.8 [0.1 to 1.4]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: There was no risk related to participating in this study as it involved implementing duties that are typically assigned to a teacher in a school.
Arm/Group | ABC for Fitness | Take 10 | GoNoodle
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/34 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/34 | 0/4
Other Adverse Events (participants affected / at risk) | 0/19 | 0/34 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT03394846/Prot_SAP_000.pdf